CLINICAL TRIAL: NCT04028323
Title: Functional MRI-based Assessment of Terlipressin vs. Octreotide on Renal Function in Cirrhotic Patients With Acute Variceal Bleeding (CHESS1903): A Multicenter, Single-blind, Randomised Controlled Trial
Brief Title: Functional MRI-based Assessment of Terlipressin vs. Octreotide on Renal Function in Cirrhotic Patients With Acute Variceal Bleeding (CHESS1903)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: LanZhou University (Other); Zhongda Hospital (Other); Guangdong Second Provincial General Hospital (Other); Xingtai People's Hospital (Other); The Third Hospital of Zhenjiang Affiliated Jiangsu University (Unknown); Tianjin Second People's Hospital (Other); The Second Hospital of Anhui Medical University (Other); The Sixth People's Hospital of Shenyang (Other); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Principal Investigator, Hepatic Hemodynamic Lab, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHESS1903
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Renal Function Disorder; Acute Variceal Bleeding
Keywords: Functional MRI; Terlipressin; Octreotide; Renal function disorder; Acute variceal bleeding
MeSH Terms: interventions — Terlipressin; Octreotide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Drug: Terlipressin. Terlipressin should be administrated with an initial dose of 1-2 mg intravenously and slowly injected (over 1 minute) while monitoring the heart rate and blood pressure. The maintenance dose should be administrated every 4-6 hours. Each dose of terlipressin is 1mg. The usual duration of therapy is 3-5 days.
  Interventions: Drug: Terlipressin
- Control group (Active Comparator): Drug: Octreotide. Octreotide should be continuously and intravenously dripped at the speed of 0.025-0.05 mg/h and could be diluted with saline with the maximum duration of 5 days. The usual duration of therapy is 3-5 days.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Terlipressin — Terlipressin should be administrated intravenously while monitoring heart rate and blood pressure daily.
  Arms: Experimental group
Drug: Octreotide — Octreotide should be continuously intravenously administrated while monitoring heart rate and blood pressure daily.
  Arms: Control group

SUMMARY:
Acute variceal bleeding is one of the critical complications in patients with cirrhosis. Due to remarkable improvements in diagnostic and therapeutic modalities such as vasoactive agents, endoscopic therapy and antibiotics, the overall prognosis has been improved during the past several decades. However, it is still associated with increased mortality that is still around 20% at 6 weeks.

Patients with advanced cirrhosis have an intense overactivity of the endogenous vasoactive systems characterized by arterial hypotension and low peripheral vascular resistance. Severe renal vasoconstriction in consequence of marked arterial vasodilatation in splanchnic circulation triggers the reduction of glomerular filtration rate, and thus induces acute kidney injury (AKI)/hepatorenal syndrome (HRS), which have been further implicated in the increasing mortality in patients with cirrhosis.

Renal functional magnetic resonance imaging (fMRI), a technique considered superior to the most common method used to estimate the glomerular filtration rate, allows for non-invasive, accurate measurements of renal structures and functions in both animals and humans. It has become increasingly prevalent in research and clinical applications. In recent years, renal fMRI has developed rapidly with progress in MRI hardware and emerging post-processing algorithms. Function related imaging markers could be acquired via renal fMRI, encompassing water molecular diffusion, perfusion, and oxygenation. The study will use phase contrast - MR angiography, intravoxel incoherent motion - diffusion weighted imaging (IVIM-DWI) and blood-oxgen-level-dependent (BOLD)-MRI to evaluate renal functional changes after using vasoactive medications in patients with cirrhosis.

The rationale for the use of vasoactive medications, including terlipressin and octreotide, is to produce splanchnic vasoconstriction and reduce portal blood flow and portal pressure, thereby underpinning the application of these vasoactive drugs in the management of cirrhotic patients with acute variceal bleeding. Meanwhile, terlipressin has been recommended as the international first-line pharmacological therapy for the treatment of HRS because terlipressin may improve renal hemodynamics, improve renal function and potentially enable HRS a reversible condition without the need of liver transplantation. However, the renal protection effect of terlipressin vs. octreotide remains unknown. In this study, the investigators aim to conduct a multicenter, single-blind randomized controlled trial to compare the renal protection effect of terlipressin vs. octreotide assessed by fMRI in the management of cirrhotic patients with acute variceal bleeding.

DETAILED DESCRIPTION:
Gastroesophageal varices, the most relevant portal-system collaterals, and acute variceal bleeding are critical complications that result directly from portal hypertension in patients with cirrhosis. Gastroesophageal varices are present approximately in 50% of patients with cirrhosis. Their presence correlates with the severity of liver disease. Only 40% of Child-Pugh A patients have varices whilst 85% of the occurrence rate in Child-Pugh C patients. Due to remarkable improvements in diagnostic and therapeutic modalities such as vasoactive agents, endoscopic therapy and antibiotics, the overall prognosis has been improved during the past several decades. However, it is still associated with increased mortality, which is still around 20% at 6 weeks. Acute variceal bleeding is also responsible for a variety of other complications in patients with cirrhosis including acute on chronic liver failure, hepatorenal syndrome, ascites liquid infection and hepatic encephalopathy. Therefore, timely and effective control of acute variceal bleeding is of crucial importance for the prognosis in patients with cirrhosis.

In the early stages of cirrhosis, when portal hypertension is moderate, increased cardiac output compensated for a modest reduction in the systemic vascular resistance, ensuring the arterial pressure and effective arterial blood volume to maintain within the normal limits. Patients with advanced cirrhosis have an intense overactivity of the endogenous vasoactive systems characterized by arterial hypotension and low peripheral vascular resistance. This cascade of events sets the stage for further renal vasoconstriction and renal sodium retention as the splanchnic and systemic vasodilatation worsens with the progression of cirrhosis. Severe renal vasoconstriction in consequence of marked arterial vasodilatation in splanchnic circulation triggers the reduction of glomerular filtration rate, and thus induces acute kidney injury (AKI)/ hepato-renal syndrome (HRS) which may implicate in the increasing mortality in patients with cirrhosis.

Renal functional magnetic resonance imaging (fMRI), a technique considered superior to the most common method used to estimate the glomerular filtration rate, allows for non-invasive, accurate measurements of renal structures and functions in both animals and humans. It has become increasingly prevalent in research and clinical applications. In recent years, renal fMRI has developed rapidly with progress in MRI hardware and emerging post-processing algorithms. Function related imaging markers could be acquired via renal fMRI, encompassing water molecular diffusion, perfusion, and oxygenation. The study will use phase contrast - MR angiography, intravoxel incoherent motion - diffusion weighted imaging (IVIM-DWI) and blood-oxgen-level-dependent (BOLD)-MRI to evaluate renal functional changes after using vasoactive medications in patients with cirrhosis.

The rationale for the use of vasoactive medications, including terlipressin and octreotide, is to produce splanchnic vasoconstriction and reduce portal blood flow and portal pressure, thereby underpinning the application of these vasoactive drugs in the management of cirrhotic patients with acute variceal bleeding. Meanwhile, terlipressin has been recommended as the international first-line pharmacological therapy for the treatment of HRS because terlipressin may improve renal hemodynamics, improve renal function in patients and potentially enable HRS a reversible condition without the need of liver transplantation. However, the renal protection effect of terlipressin vs. octreotide remains unknown. In this study, the investigators aim to conduct a multicenter, single-blind randomized controlled trial to compare the renal protection effect of terlipressin vs. octreotide assessed by fMRI in the management of cirrhotic patients with acute variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* clinically and/or pathologically diagnosed cirrhosis
* with a clinical history of acute variceal bleeding (melena, hematemesis etc.) assessed as Child-Pugh class B or C
* voluntarily participated in the study and able to provide written informed consent and able to understand and willing to comply with the requirements of the study

Exclusion Criteria:

* pregnant or lactating woman
* diagnosed or suspected malignancy (hepatocellular carcinoma, cholangiocarcinoma etc.)
* with mental disease and unable to comply with MRI examination
* with contraindications of terlipressin and octreotide
* with other conditions judged inadequate for participation by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Renal function | 6 days
  Number of participants with the improvement of renal function assessed by serum creatinine

SECONDARY OUTCOMES:
Renal perfusion | 6 days
  Number of participants with the improvement of renal perfusion assessed by functional MRI measurement (intravoxel incoherent motion)
Renal blood oxygenation | 6 days
  Number of participants with the improvement of renal blood oxygenation assessed by functional MRI measurement (blood oxygen level dependent)
Failure to control bleeding | 6 days
  The occurrence rate of failure to control bleeding
Intra-hospital rebleeding | 6 days
  The occurrence rate of intra-hospital rebleeding
Intra-hospital mortality | 6 days
  The occurrence rate of intra-hospital mortality
Adverse events | 6 days
  The occurrence rate of adverse events
Overall survival | 90 days
  The number of participants still alive with the 90 days follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shenghong Ju, MD, Principal Investigator — Zhongda Hospital; Xingshun Qi, MD, Principal Investigator — General Hospital of Shenyang Military Area; Xiaolong Qi, MD, Principal Investigator — LanZhou University
Locations (10):
- China (10):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - Zhongda Hospital, Medical School, Southeast University, Nanjing, Jiangsu
  - The Third Hospital of Zhenjiang Affiliated Jiangsu University, Zhenjiang, Jiangsu
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - The Second Affiliated Hospital of Baotou Medical University, Baotou, Neimenggu
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gines P, Schrier RW. Renal failure in cirrhosis. N Engl J Med. 2009 Sep 24;361(13):1279-90. doi: 10.1056/NEJMra0809139. No abstract available. PMID 19776409
- [Background] Ibrahim M, Mostafa I, Deviere J. New Developments in Managing Variceal Bleeding. Gastroenterology. 2018 May;154(7):1964-1969. doi: 10.1053/j.gastro.2018.02.023. Epub 2018 Mar 2. PMID 29481777
- [Background] Wong F. Recent advances in our understanding of hepatorenal syndrome. Nat Rev Gastroenterol Hepatol. 2012 May 22;9(7):382-91. doi: 10.1038/nrgastro.2012.96. PMID 22614754
- [Background] Martin-Llahi M, Pepin MN, Guevara M, Diaz F, Torre A, Monescillo A, Soriano G, Terra C, Fabrega E, Arroyo V, Rodes J, Gines P; TAHRS Investigators. Terlipressin and albumin vs albumin in patients with cirrhosis and hepatorenal syndrome: a randomized study. Gastroenterology. 2008 May;134(5):1352-9. doi: 10.1053/j.gastro.2008.02.024. Epub 2008 Feb 14. PMID 18471512
- [Background] Levacher S, Letoumelin P, Pateron D, Blaise M, Lapandry C, Pourriat JL. Early administration of terlipressin plus glyceryl trinitrate to control active upper gastrointestinal bleeding in cirrhotic patients. Lancet. 1995 Sep 30;346(8979):865-8. doi: 10.1016/s0140-6736(95)92708-5. PMID 7564670
- [Background] Seo YS, Park SY, Kim MY, Kim JH, Park JY, Yim HJ, Jang BK, Kim HS, Hahn T, Kim BI, Heo J, An H, Tak WY, Baik SK, Han KH, Hwang JS, Park SH, Cho M, Um SH. Lack of difference among terlipressin, somatostatin, and octreotide in the control of acute gastroesophageal variceal hemorrhage. Hepatology. 2014 Sep;60(3):954-63. doi: 10.1002/hep.27006. Epub 2014 Jul 25. PMID 24415445
- [Background] Abid S, Jafri W, Hamid S, Salih M, Azam Z, Mumtaz K, Shah HA, Abbas Z. Terlipressin vs. octreotide in bleeding esophageal varices as an adjuvant therapy with endoscopic band ligation: a randomized double-blind placebo-controlled trial. Am J Gastroenterol. 2009 Mar;104(3):617-23. doi: 10.1038/ajg.2008.147. Epub 2009 Feb 17. PMID 19223890
- [Background] Cavallin M, Kamath PS, Merli M, Fasolato S, Toniutto P, Salerno F, Bernardi M, Romanelli RG, Colletta C, Salinas F, Di Giacomo A, Ridola L, Fornasiere E, Caraceni P, Morando F, Piano S, Gatta A, Angeli P; Italian Association for the Study of the Liver Study Group on Hepatorenal Syndrome. Terlipressin plus albumin versus midodrine and octreotide plus albumin in the treatment of hepatorenal syndrome: A randomized trial. Hepatology. 2015 Aug;62(2):567-74. doi: 10.1002/hep.27709. Epub 2015 Feb 13. PMID 25644760
- [Background] Wang YC, Tang A, Chang D, Zhang SJ, Ju S. Significant perturbation in renal functional magnetic resonance imaging parameters and contrast retention for iodixanol compared with iopromide: an experimental study using blood-oxygen-level-dependent/diffusion-weighted magnetic resonance imaging and computed tomography in rats. Invest Radiol. 2014 Nov;49(11):699-706. doi: 10.1097/RLI.0000000000000073. PMID 24879299
- [Background] Chang D, Wang YC, Xu TT, Peng XG, Cai Y, Wang L, Bai YY, Ju S. Noninvasive Identification of Renal Hypoxia in Experimental Myocardial Infarctions of Different Sizes by Using BOLD MR Imaging in a Mouse Model. Radiology. 2018 Jan;286(1):129-139. doi: 10.1148/radiol.2017161998. Epub 2017 Aug 4. PMID 28777704
- [Derived] Yan X, Shao R, Wang Y, Mao X, Lei J, Zhang L, Zheng J, Liu A, Zhao H, Gao F, Wang J, Li P, Yao S, Xu M, Xu J, Liu D, Mi Y, Gong X, Ye J, Deng M, Dang T, Ji J, Shao C, Liu C, Gu Y, Wu Y, Wang F, Teng G, Li X, Qi X, Ju S, Qi X. Functional magnetic resonance imaging-based assessment of terlipressin vs. octreotide on renal function in cirrhotic patients with acute variceal bleeding (CHESS1903): study protocol of a multicenter randomized controlled trial. Ann Transl Med. 2019 Oct;7(20):586. doi: 10.21037/atm.2019.09.141. PMID 31807567